CLINICAL TRIAL: NCT05541224
Title: A Retrospective Epidemiologic Registry to Gain Insight Into the Characteristics and Prognosis of AML Patients According to the Routinely Used Genetic and Biologic Markers
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: REAL-MOL
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: De novo Acute Myeloid Leukemia; Relapsed/refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, translational, epidemiologic, multicenter, non-interventional study (No EPA study) to provide insights into disease epidemiology, disease biology, treatment regimens, and clinical outcomes of patients with acute myeloblastic leukemia (AML) in routine clinical practice according to their molecular markers.

The primary objective of the study is to describe the use of the main molecular markers (FLT3 and NPM1) in the real-life according of the type of AML, treating institution, patients' characteristics, and disease status.

DETAILED DESCRIPTION:
This is a retrospective, translational, epidemiologic, multicenter, non-interventional study (No EPA study) to provide insights into disease epidemiology, disease biology, treatment regimens, and clinical outcomes of patients with AML in routine clinical practice according to their molecular markers.

Once it has been confirmed that all selection criteria for the study have been met and informed consent has been obtained, the subject will be considered enrolled in the study and the investigator can proceed to collect data from their medical record by completing a case report (CRF).

The study contemplates the retrospective collection of data from disease diagnosis to the start of the study. Only data obtained before the start of the study will be collected in order to ensure they are retrospective in nature.

The study will be conducted following the requirements contained in the Declaration of Helsinki (Fortaleza, Brazil 2013) and in accordance with the current Spanish legislation with regard to conducting observational studies (Ministerial Order SAS/3470/2009).

The primary objective of the study is to describe the use of the main molecular markers (FLT3 and NPM1) in the real-life according of the type of AML, treating institution, patients' characteristics, and disease status.

This project will be conducted in the Spanish PETHEMA cooperative group, constituted by 60 institutions and seven main central laboratories with extensive technological capacity. All patients will be included in the ongoing PETHEMA epidemiologic registry of AML with the purpose to collect a large number, additional and non-pre-existent clinical data, including first-line and salvage treatment schedules and outcomes of each patient.

For this study the PETHEMA AML registry will be enlarged seeking for new cases not previously reported. The data base information will be updated emphasizing for the capture of new data on molecular screening tests performed on a routine basis (FLT3, NPM1, and others). For these purpose, information will be systematically requested from the main PETHEMA laboratories. Therapies and clinical outcome data will be retrospectively collected. This is a one-step study without intervention, in which all analyses will be performed at the end of the database completion.

ELIGIBILITY:
Inclusion Criteria:

1. All adult patients with AML (excluding APL) according to the WHO criteria (2008), regardless of the treatment administered by their treating physician.
2. AML at diagnosis and at relapse or refractoriness.
3. Patients from institutions participating in the ongoing PETHEMA AML registry.
4. Patients with information about the molecular screening including FLT3 with or without NPM1 mutations (including positive/negative or not performed).
5. Ability to give informed consent before the study initiation. Death patients and patients who are no longer contactable or lost to follow-up will be excluded from consent requirement.

Exclusion Criteria:

1. Pediatric patients.
2. Acute promyelocytic leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with AML (new diagnosis or relapsed/refractory disease). These patients must meet all the inclusion criteria and none of the exclusion criteria specified.
Sampling Method: Non-Probability Sample
Enrollment: 6917 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with molecular alterations (FLT3 and NPM1 mutations). | Baseline
  Percentage of each of the standard screening panel molecular alterations studied in the AML patients (FLT3 and NPM1) by AML type, by center, by patient's characteristics and the disease status.

SECONDARY OUTCOMES:
Overall response rate. | Throughout the study period. Approximately 1 year
  Percentage of patients achieving response in each group of the baseline alterations studied in the AML patients (FLT3 and NPM1) .
Description of initial and later treatments in each baseline alterations studied (FLT3 and NPM1) in each AML type. | Baseline and throughout the study period. Approximately 1 year
  Frequency of initial and later type of treatments in each baseline alterations studied (FLT3 and NPM1) in each AML type.
Molecular response rate. | Throughout the study period. Approximately 1 year
  Percentage of patients achieving molecular response in each group of the baseline alterations studied in the AML patients (FLT3 and NPM1) .
Description of biology of disease at relapse or refractoriness by molecular characteristics. | Baseline and throughout the study period. Approximately 1 year
  Percentage of AML type at relapse or refractoriness in each baseline alterations studied (FLT3 and NPM1).

CONTACTS AND LOCATIONS:
Overall Officials: Pau Montesinos Fernández, Study Chair — Hospital Universitari i Politècnic La Fe (Valencia)
Locations (22):
- Spain (22):
  - Hospital General Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Germans Trias i Pujol-ICO, Badalona
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario de Castellón, Castellon
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Univeristario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central Asturias, Oviedo
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari I Politécnic La Fe, Valencia
  - Hospital Universitario Doctor Peset, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schlenk RF, Dohner K, Krauter J, Frohling S, Corbacioglu A, Bullinger L, Habdank M, Spath D, Morgan M, Benner A, Schlegelberger B, Heil G, Ganser A, Dohner H; German-Austrian Acute Myeloid Leukemia Study Group. Mutations and treatment outcome in cytogenetically normal acute myeloid leukemia. N Engl J Med. 2008 May 1;358(18):1909-18. doi: 10.1056/NEJMoa074306. PMID 18450602
- [Background] Thiede C, Steudel C, Mohr B, Schaich M, Schakel U, Platzbecker U, Wermke M, Bornhauser M, Ritter M, Neubauer A, Ehninger G, Illmer T. Analysis of FLT3-activating mutations in 979 patients with acute myelogenous leukemia: association with FAB subtypes and identification of subgroups with poor prognosis. Blood. 2002 Jun 15;99(12):4326-35. doi: 10.1182/blood.v99.12.4326. PMID 12036858
- [Background] Frohling S, Schlenk RF, Breitruck J, Benner A, Kreitmeier S, Tobis K, Dohner H, Dohner K; AML Study Group Ulm. Acute myeloid leukemia. Prognostic significance of activating FLT3 mutations in younger adults (16 to 60 years) with acute myeloid leukemia and normal cytogenetics: a study of the AML Study Group Ulm. Blood. 2002 Dec 15;100(13):4372-80. doi: 10.1182/blood-2002-05-1440. Epub 2002 Aug 8. PMID 12393388
- [Background] Kottaridis PD, Gale RE, Frew ME, Harrison G, Langabeer SE, Belton AA, Walker H, Wheatley K, Bowen DT, Burnett AK, Goldstone AH, Linch DC. The presence of a FLT3 internal tandem duplication in patients with acute myeloid leukemia (AML) adds important prognostic information to cytogenetic risk group and response to the first cycle of chemotherapy: analysis of 854 patients from the United Kingdom Medical Research Council AML 10 and 12 trials. Blood. 2001 Sep 15;98(6):1752-9. doi: 10.1182/blood.v98.6.1752. PMID 11535508
- [Background] Gale RE, Hills R, Kottaridis PD, Srirangan S, Wheatley K, Burnett AK, Linch DC. No evidence that FLT3 status should be considered as an indicator for transplantation in acute myeloid leukemia (AML): an analysis of 1135 patients, excluding acute promyelocytic leukemia, from the UK MRC AML10 and 12 trials. Blood. 2005 Nov 15;106(10):3658-65. doi: 10.1182/blood-2005-03-1323. Epub 2005 Aug 2. PMID 16076872
- [Background] Rombouts WJ, Blokland I, Lowenberg B, Ploemacher RE. Biological characteristics and prognosis of adult acute myeloid leukemia with internal tandem duplications in the Flt3 gene. Leukemia. 2000 Apr;14(4):675-83. doi: 10.1038/sj.leu.2401731. PMID 10764154
- [Background] Yokota S, Kiyoi H, Nakao M, Iwai T, Misawa S, Okuda T, Sonoda Y, Abe T, Kahsima K, Matsuo Y, Naoe T. Internal tandem duplication of the FLT3 gene is preferentially seen in acute myeloid leukemia and myelodysplastic syndrome among various hematological malignancies. A study on a large series of patients and cell lines. Leukemia. 1997 Oct;11(10):1605-9. doi: 10.1038/sj.leu.2400812. PMID 9324277
- [Background] Whitman SP, Archer KJ, Feng L, Baldus C, Becknell B, Carlson BD, Carroll AJ, Mrozek K, Vardiman JW, George SL, Kolitz JE, Larson RA, Bloomfield CD, Caligiuri MA. Absence of the wild-type allele predicts poor prognosis in adult de novo acute myeloid leukemia with normal cytogenetics and the internal tandem duplication of FLT3: a cancer and leukemia group B study. Cancer Res. 2001 Oct 1;61(19):7233-9. PMID 11585760
- [Background] Dohner K, Schlenk RF, Habdank M, Scholl C, Rucker FG, Corbacioglu A, Bullinger L, Frohling S, Dohner H. Mutant nucleophosmin (NPM1) predicts favorable prognosis in younger adults with acute myeloid leukemia and normal cytogenetics: interaction with other gene mutations. Blood. 2005 Dec 1;106(12):3740-6. doi: 10.1182/blood-2005-05-2164. Epub 2005 Jul 28. PMID 16051734
- [Background] Verhaak RG, Goudswaard CS, van Putten W, Bijl MA, Sanders MA, Hugens W, Uitterlinden AG, Erpelinck CA, Delwel R, Lowenberg B, Valk PJ. Mutations in nucleophosmin (NPM1) in acute myeloid leukemia (AML): association with other gene abnormalities and previously established gene expression signatures and their favorable prognostic significance. Blood. 2005 Dec 1;106(12):3747-54. doi: 10.1182/blood-2005-05-2168. Epub 2005 Aug 18. PMID 16109776
- [Background] Suzuki T, Kiyoi H, Ozeki K, Tomita A, Yamaji S, Suzuki R, Kodera Y, Miyawaki S, Asou N, Kuriyama K, Yagasaki F, Shimazaki C, Akiyama H, Nishimura M, Motoji T, Shinagawa K, Takeshita A, Ueda R, Kinoshita T, Emi N, Naoe T. Clinical characteristics and prognostic implications of NPM1 mutations in acute myeloid leukemia. Blood. 2005 Oct 15;106(8):2854-61. doi: 10.1182/blood-2005-04-1733. Epub 2005 Jun 30. PMID 15994285
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Hellmann F, Verdi M, Schlemper BR Jr, Caponi S. 50th anniversary of the Declaration of Helsinki: the double standard was introduced. Arch Med Res. 2014 Oct;45(7):600-1. doi: 10.1016/j.arcmed.2014.10.005. Epub 2014 Oct 31. PMID 25450586